CLINICAL TRIAL: NCT00335114
Title: Efficacy of Cyclosporine Ophthalmic Emulsion in the Treatment of Dry Eye Syndrome in Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Carol E. Rosenstiel, Professor, Director of Contact Lens Service, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F051025017
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Contact Lens Wearers With Dry Eye Syndrome
Keywords: cyclosporine, dry eye syndrome, contact lens
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion

SUMMARY:
Cyclosporine Ophthalmic Emulsion is currently used in the treatment of dry eye syndrome. Contact lens wearers frequently suffer from dry eye syndrome. The purpose of this study is to evaluate cyclosporine ophthalmic emulsion verses re-wetting drops in the relief of dry eye symptoms in contact lens wearers

ELIGIBILITY:
Inclusion Criteria:

* contact lens wearer
* clinical diagnosis of dry eye syndrome

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Ocular exams and questionnaires at baseline and at 3 months will determine
the effect of cyclosporine on dry eye syndrome.

SECONDARY OUTCOMES:
Increased contact lens wearing time due to a decrease in severity
of dry eye symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Carol E Rosenstiel, OD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Ophthalmology Services Foundation, Birmingham, Alabama, United States